CLINICAL TRIAL: NCT00923299
Title: Phase I-II Study Evaluating Combined Treatment of Cetuximab and Trastuzumab in Metastatic Pancreatic Cancer Patients Progressing After Gemcitabine Based Chemotherapy.(THERAPY)
Brief Title: Cetuximab and Trastuzumab in Treating Patients With Metastatic Pancreatic Cancer That Progressed After Previous Treatment With Gemcitabine
Acronym: THERAPY
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000636018; CLCC-THERAPY; RECF0910; VA-2008/34; EUDRACT-2008-003988-39
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Cancer
Keywords: stage IV pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cetuximab, trastuzumab (Other)
  Interventions: Drug: cetuximab; Drug: trastuzumab

INTERVENTIONS:
Drug: cetuximab — Cetuximab at the initial dose of 400 mg/m² (J1S1) as a 2-hour infusion and then at the 250 mg/m² dose as a 1-hour infusion in subsequent weeks.
Drug: trastuzumab — Two dose levels of trastuzumab will be evaluated for Phase 1:
  * Level 1: a loading dose of 3 mg/kg as a 90-minute intravenous infusion at J1S1 and then 1.5 mg/kg as a 30-minute intravenous infusion for all subsequent weekly administrations;
  * Level 2: a loading dose of 4 mg/kg as a 90-minute intravenous infusion at J1S1 and then 2 mg/kg as a 30-minute intravenous infusion for all subsequent weekly administrations.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab and trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving cetuximab together with trastuzumab may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of trastuzumab when given together with cetuximab and to see how well it works in treating patients with metastatic pancreatic cancer that progressed after previous treatment with gemcitabine.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the recommended dose of trastuzumab when given with cetuximab in patients with metastatic pancreatic cancer that progressed after gemcitabine-based chemotherapy. (Phase I)
* Evaluate the objective response rate as assessed by RECIST criteria. (Phase II)

Secondary

* Evaluate the safety profile as assessed by NCI CTCAE v3.0.
* Evaluate progression-free survival.
* Evaluate overall survival.

OUTLINE: This is a multicenter, phase I dose-escalation study of trastuzumab followed by a phase II study.

Patients receive cetuximab IV over 1-2 hours and trastuzumab IV over 30-90 minutes on day 1. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic adenocarcinoma of the pancreas

  * Progressed after first-line or adjuvant gemcitabine-based chemotherapy
* Measurable disease as assessed by RECIST criteria
* No known brain metastasis or symptomatic carcinomatous leptomeningitis

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy ≥ 3 months
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 2.5 times ULN
* ALT/AST ≤ 5 times ULN
* LVEF ≥ 55%
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No significant comorbidities, including any of the following:

  * Cardiovascular disease
  * Documented history of congestive heart failure
  * Uncontrolled, high-risk arrhythmia
  * Angina pectoris requiring treatment
  * Clinically significant valvular disease
  * Evidence of transmural myocardial infarction by ECG
  * Uncontrolled hypertension
  * Active bleeding
  * Clinically significant active infection
  * Severe dyspnea at rest
  * Oxygen-dependency
* No other malignancy except basal cell carcinoma of the skin
* No severe hypersensitivity to cetuximab or trastuzumab
* No medical or psychological condition that would preclude study completion or giving informed consent
* No legal incapacity or limited legal capacity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior cetuximab or trastuzumab
* No other concurrent experimental drugs or anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Recommended dose of trastuzumab when given with cetuximab (Phase I) | 15 days
  From baseline to the end of treatment
Objective response rate as assessed by RECIST criteria (Phase II) | Approximately 8 weeks
  From baseline to the end of treatment

SECONDARY OUTCOMES:
Progression-free survival | Approximately 36 months
  From baseline to the end of study
Overall survival | Approximately 36 months
  From baseline to the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ychou, MD, PhD, Principal Investigator — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France

REFERENCES:
- [Result] Assenat E, Azria D, Mollevi C, Guimbaud R, Tubiana-Mathieu N, Smith D, Delord JP, Samalin E, Portales F, Larbouret C, Robert B, Bibeau F, Bleuse JP, Crapez E, Ychou M, Pelegrin A. Dual targeting of HER1/EGFR and HER2 with cetuximab and trastuzumab in patients with metastatic pancreatic cancer after gemcitabine failure: results of the "THERAPY"phase 1-2 trial. Oncotarget. 2015 May 20;6(14):12796-808. doi: 10.18632/oncotarget.3473. PMID 25918250